CLINICAL TRIAL: NCT02054065
Title: Effect of CAUTI Prevention Alert - A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12-06-225
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Infection Due to Indwelling Urinary Catheter
Keywords: Urinary Catheter; urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Normal care conditions, no computer-based physician alert.
- CAUTI Decision Support (Experimental): Decision support aimed at preventing Catheter Associated Urinary Tract Infections (CAUTIs)
  Interventions: Other: CAUTI Decision Support

INTERVENTIONS:
Other: CAUTI Decision Support — Decision support used to prevent Catheter Associated Urinary Tract Infections
  Arms: CAUTI Decision Support

SUMMARY:
This study proposes to expand upon previous research by studying the effects of a urinary-catheter removal alert on duration of urinary catheter use and frequency of CAUTIs with a large, randomized controlled trial within a three-hospital academic medical center.

Hypothesis The proposed urinary-catheter removal alerts will decrease the number of catheter days and decrease the number of catheter associated urinary tract infections (CAUTIs), but will not affect the catheter re-insertion rate.

DETAILED DESCRIPTION:
Primary Objectives

* Specific Aim 1: Investigate the effect of a urinary-catheter removal alert on the rate of catheter associated urinary tract infections (CAUTIs).
* Specific Aim 2: Investigate the effect of a urinary-catheter removal alert on the number of catheter days.
* Specific Aim 3: Evaluate the effect of a urinary-catheter removal alert on the rate of catheter re-insertion.
* Specific Aim 4: Evaluate the effect of a urinary-catheter removal alert on overall mortality in patients with indwelling catheters.

ELIGIBILITY:
Inclusion Criteria:

* All admissions with an indwelling urinary catheter will be randomly assigned to intervention vs. control (usual care) conditions.

Exclusion Criteria:

* Neonatal Intensive Care Unit and pediatric patients

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of CAUTIs | One Year

SECONDARY OUTCOMES:
Number of catheter days | One year
Rate of catheter re-insertion | One Year
Patient mortality due to CAUTI | One year

CONTACTS AND LOCATIONS:
Overall Officials: Jason S Adelman, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, New York, New York, United States